CLINICAL TRIAL: NCT01919203
Title: the Effective Bolus Dose of Remifentanil for Laryngeal Mask Airway (LMA) Insertion in Pediatric Patients
Brief Title: the Effective Bolus Dose of Remifentanil for Laryngeal Mask Airway (LMA) Insertion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangjin Park (Other)
Responsible Party: Sponsor-Investigator, Sangjin Park, assistant professor, Yeungnam University College of Medicine
Organization: Yeungnam University College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: apsj0723
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Complication
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- group R (Experimental): The starting dose of remifentanil is 0.5μg/kg and a step size was 0.05μg/kg.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — The starting dose of remifentanil is 0.5μg/kg and a step size is 0.05μg/kg. If LMA insertion is successful or failed in previous patient, an decrement or increment of 0.05μg/kg remifentanil is injected to next patient, respectively.
  Other Names: remifentanil (ultiva)

SUMMARY:
This research attempts to find the optimum dose of remifentanil that can prevent the unnecessary responses such as coughing, gagging, and movement when LMA is inserted during sevoflurane induction in pediatric patients.

DETAILED DESCRIPTION:
Anaesthesia is induced by inhalation with 3% sevoflurane. A predetermined bolus dose of remifentanil is injected over 30 seconds. The LMA is attempted 60 seconds after bolus administration. The starting dose of remifentanil is 0.5μg/kg and a step size is 0.05μg/kg. If LMA insertion is successful or failed in previous patient, an decrement or increment of 0.05μg/kg remifentanil is injected to next patient, respectively.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1 or 2
* undergoing short elective surgery(i.e Strabismus surgery, Entropion surgery, Inguinal hernia surgery, etc) under general anesthesia

Exclusion Criteria:

* suspected difficult airways
* respiratory disease (chronic obstructive pulmonary disease, upper respiratory infection)
* body mass index > 30 kg/m2
* allergies to the study drugs
* a history of gastric reflux

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
patients's response to the LMA insertion | 2 minutes after LMA insertion
  Fail of LMA insertion is defined as body or limb movement, coughing or gagging with 2 minutes after LMA insertion, no proper jaw relaxation(difficult mouth opening), laryngospasm, bronchospasm, desaturation(SpO2<94%)

CONTACTS AND LOCATIONS:
Overall Officials: sangjin park, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, College of medicine, Yeungnam University, Daemyung-Dong, Nam-Gu, Daegu, Republic of Korea
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yeungnam University hospital, Nam Gu, Daegu, South Korea